CLINICAL TRIAL: NCT00274638
Title: A Prospective, Randomised, Open-Label, Blinded-Endpoint, Parallel Group 6-week Treatment Study Comparing Telmisartan Combined With Hydrochlorothiazide (40 mg/12.5 mg or 80 mg/12.5 mg) Tablets With Losartan Combined With Hydrochlorothiazide (50 mg/12.5 mg) Tablets Using Ambulatory Blood Pressure Monitoring in Patients With Mild-to-Moderate Hypertension
Brief Title: PROBE Parallel 6-week Treatment Comparing Telmisartan/Hydrochlorothiazide (HCT) (40/12.5 or 80/12.5) With Losartan/HCT (50/12.5) Using Ambulatory Blood Pressure Monitoring (ABPM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 502.387
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — telmisartan, hydrochlorothiazide drug combination; hydrochlorothiazide, losartan drug combination

INTERVENTIONS:
Drug: Telmisartan & Hydrochlorothiazide
Drug: Losartan & Hydrochlorothiazide
Procedure: ABPM

SUMMARY:
To demonstrate that Telmisartan combined with Hydrochlorothiazide (MICARDIS® HCT) is superior to Losartan with Hydrochlorothiazide (Hyzaar®) in lowering blood pressure in mild-moderate hypertensives.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent in accordance with GCP and local legislation.
2. Mild-to-moderate hypertension defined as a mean seated DBP of >= 95 mm Hg and <=l to 109 mm Hg, measured by manual cuff sphygmomanometer at Visit 2.
3. Male or Female >= 18 years.
4. Ability to stop any current antihypertensive therapy without risk to the patient (investigator's discretion).
5. 24-hour ABPM mean DBP of >= 85 mm Hg at Visit 3.

Exclusion Criteria:

1. Pre-menopausal women (last menstruation <= 1 year prior to signing informed consent) who

   * are not surgically sterile, or are
   * nursing, or
   * are of child-bearing potential and are NOT practicing acceptable methods of birth control, or do not plan to continue practicing an acceptable method throughout the study. Acceptable methods of birth control include IUD, oral, implantable or injectable contraceptives. No exception will be made.
2. Night shift workers who routinely sleep during the daytime and whose work hours include midnight to 4:00 A.M.
3. Mean seated SBP >= 180 mm Hg or mean seated DBP >= 110 mm Hg during any visit or the placebo run-in phase.
4. Known or suspected secondary hypertension (i.e. pheochromocytoma).
5. Hepatic and/or renal dysfunction as defined by the following laboratory parameters: a)SGPT (ALT) or (SGOT) AST less than two times the upper limit of normal range, or b)Serum creatinine greater than 2.3 mg/dL (>203 mico mol/l).
6. Bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, post-renal transplant patients or patients with only one kidney.
7. Biliary obstructive disorders.
8. Clinically relevant sodium depletion, hypokalaemia or hyperkalaemia.
9. Uncorrected volume depletion.
10. Primary aldosteronism.
11. Hereditary fructose intolerance.
12. Congestive heart failure (NYHA functional class CHF III-IV).
13. Unstable angina within the past 3 months prior to signing the informed consent form.
14. Stroke within the past 6 months prior to signing the informed consent form.
15. Myocardial infarction or cardiac surgery within the past 3 months prior to signing the inform consent form.
16. PTCA (percutaneous transluminal coronary angioplasty) within the past 3 months prior to signing the informed consent form.
17. Sustained ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the investigator.
18. Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of the aortic or mitral valve.
19. Patients with insulin-dependent diabetes mellitus whose diabetes has not been stable and controlled for at least the past 3 months as defined by an HbA1C >= 10 Percent.
20. Patients who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or angiotensin II receptor antagonists.
21. History of drug or alcohol dependency within 6 months prior to signing the informed consent form.
22. Chronic administration of any medications known to affect blood pressure, except medication allowed by the protocol.
23. Any investigational therapy within 1 month of signing the informed consent form.
24. Known hypersensitivity to any component of the study drugs (placebo, telmisartan, hydrochlorothiazide or losartan).
25. Any clinical condition which, in the opinion of the investigator would not allow safe completion of the protocol and safe administration of trial medication.
26. Concomitant use of lithium or cholestyramine or colestipol resins (potential drug interactions with hydrochlorothiazide).
27. History of non-compliance with prescribed medication.
28. Inability to comply with protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 805 (Actual)
Dates: Start 2002-07; Primary Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the last 6-hour mean (relative to dose time) diastolic blood pressure (DBP) as measured by ABPM (Ambulatory Blood Pressure Monitoring) | after 6 Weeks

SECONDARY OUTCOMES:
Change in the last 6-hour ABPM mean (relative to dosing time) for systolic blood pressure (SBP) | after 6 weeks
Change in the 24-hour ABPM mean (relative to dosing time) for DBP and SBP | after 6 weeks
Change in the ABPM mean DBP and SBP during the morning, daytime, and night-time periods of the 24-hour dosing interval | after 6 weeks
Change in systolic and diastolic blood pressure load during the 24-hour dosing interval of the 24-hour dosing interval | after 6 weeks
Change in mean seated trough DBP and SBP as measured by manual in-clinic cuff sphygmomanometer | after 6 weeks
Responder rates based on both the 24-hour ABPM mean (relative to dose time) blood pressures and the in-clinic trough cuff measurements | after 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (69):
- United States (69):
  - Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - Research Solutions, LLC, Little Rock, Arkansas
  - Boehringer Ingelheim Investigational Site, Carmichael, California
  - Boehringer Ingelheim Investigational Site, Concord, California
  - Sierra Medical Research, Fresno, California
  - Attn: Ginger Paselk, Long Beach, California
  - Boehringer Ingelheim Investigational Site, Orange, California
  - DeBruin Medical Center, Orangevale, California
  - Clinical Trials Research, Roseville, California
  - Dr. R. David Ferrera, Sacramento, California
  - Westlake Medical Research, Westlake Village, California
  - Rocky Mountain Pulmonary & Critical Care Medicine, Inc., Wheat Ridge, Colorado
  - Clinical Research Consultants, Inc., Trumbull, Connecticut
  - Glasgow Family Pract6ice, Newark, Delaware
  - Boehringer Ingelheim Investigational Site, Coral Gables, Florida
  - Miami Research Associates, Coral Gables, Florida
  - Patron, Andres, D.O., Hollywood, Florida
  - Christopher Chappel, MD, Kissimmee, Florida
  - Boehringer Ingelheim Investigational Site, Melbourne, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Attention: Larry I. Gilderman, D.O., Pembroke Pines, Florida
  - nTouch Research, St. Petersburg, Florida
  - Tampa Medical Research Associates, Tampa, Florida
  - Southern Clinical Research and Management, Inc., Augusta, Georgia
  - Boehringer Ingelheim Investigational Site, Conyers, Georgia
  - Treasure Valley Cardiology, Boise, Idaho
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Herron Medical Center, Ltd., Chicago, Illinois
  - Protococare Trials, Inc., Elk Grove Village, Illinois
  - N Touch Research, Peoria, Illinois
  - Midwest Institute for Clinical Research Inc., Indianapolis, Indiana
  - Radiant Research, Overland, Kansas
  - Ong Medical Center, Oxon Hill, Maryland
  - Radiant Research, Edina, Minnesota
  - Cardiology Research, Saint Paul, Minnesota
  - Attention: Mel E. Lucas, DO, Florissant, Missouri
  - New Mexico Clinical Reaearch & Osteoporosis Center, Inc., Albuquerque, New Mexico
  - Syracuse Preventative Cardiology, Syracuse, New York
  - Great Lakes Medical Research, Westfield, New York
  - Cardiology and Internal Medicine- Williamsville NY, Williamsville, New York
  - Comprehensive Clinical Research, Bina, North Carolina
  - Bennett Cardiac Center, Charlotte, North Carolina
  - Charlotte Clinical Research, Charlotte, North Carolina
  - Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - nTouch Research Corporation, Raleigh, North Carolina
  - Piedmont Research Associates, Winston-Salem, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - Radiant Reseach, Cincinnati, Ohio
  - Radiant Research, Columbus, Ohio
  - Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - nTouch, Oklahoma City, Oklahoma
  - Hillcrest Medical Center, Tulsa, Oklahoma
  - Bock Clinical Research, Collegeville, Pennsylvania
  - Bock Clinical Research, Downingtown, Pennsylvania
  - Bock Clinical Research, Harleysville, Pennsylvania
  - The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Omega Research, Warwick, Rhode Island
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Veterans Affairs Medical Center, Memphis, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Boehringer Ingelheim Investigational Site, Dallas, Texas
  - nTouch Research, Houston, Texas
  - Hampton Roads Medical Specialists, Hampton, Virginia
  - 885 Kempsville Road, Suite 221, Norfolk, Virginia
  - York Clinical Research, Norfolk, Virginia
  - Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - Gemini Scientific, Madison, Wisconsin
  - University of Wisconsin Medical School, Madison, Wisconsin